CLINICAL TRIAL: NCT01508221
Title: A Phase II Trial to Evaluate the Use of Trental and Vitamin E for Prophylaxis of Radiation Necrosis
Brief Title: Evaluation of the Use of Trental and Vitamin E For Prophylaxis of Radiation Necrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michelle Marcum, Director, University of Cincinnati Cancer Center, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BTC-W1
Record Dates: First submitted 2012-01-08; First posted 2012-01-11 (Estimated); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Brain Metastasis
Keywords: brain metastasis
MeSH Terms: conditions — Brain Neoplasms | interventions — Pentoxifylline; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trental + Vitamin E (Experimental): Trental 400 mg TID and Vitamin E 400IU BID starting the first day after the last radiosurgery treatment
  Interventions: Drug: Trental; Dietary Supplement: Vitamin E

INTERVENTIONS:
Drug: Trental — 400 mg tid starting first day after last radiosurgery treatment and continuing for 6 months
  Other Names: Pentoxifylline
Dietary Supplement: Vitamin E — 400IU twice daily starting the first day after last radiosurgery treatment and continuing for 6 months

SUMMARY:
The purpose of this study is to determine whether the use of Trental and Vitamin E can help reduce the incidence of radiation necrosis (a lesion that usually occurs at the original tumor site) after radiosurgery. These two drugs are commonly used to treat radiation necrosis when it occurs but the hope is that these drugs can be used to prevent radiation necrosis from ever occurring.

DETAILED DESCRIPTION:
The treatment phase of the study is 6 months. Study procedures will be conducted such as: history, physical and neurological exam, pregnancy testing (for women of child bearing age) and a Brain MRI. Follow-up appointments will be every 3 months for 1 year at which time, your participation in the study will be concluded.

ELIGIBILITY:
Inclusion Criteria:

* Plan to undergo single or five fraction radiosurgery for a metastatic brain tumor
* Diagnosis of a metastatic brain tumor may be accomplished by histologic confirmation or by clinical confirmation by the treating physician based on MR imaging characteristics in the setting of a known history of cancer
* Age > 18 years
* Partial or total resection of a metastatic tumor are eligible

Exclusion Criteria:

* Known sensitivity to vitamin E or Trental
* Recent intracranial bleed or retinal hemorrhage
* Treatment with a non-approved or investigational drug within 30 days before day 1 of study treatment
* History of Avastin treatment
* Anticipated need for treatment with Avastin
* History of bleeding disorder
* History of liver disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Warnick, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trental + Vitamin E
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trental + Vitamin E
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 56.87 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Radiation Necrosis
Description: Number of symptomatic death of healthy tissue caused by radiation therapy.
Time Frame: average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Trental + Vitamin E
Number analyzed (Participants) | 31
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse Event collection is not specifically mapped out per protocol. The length of the study is 3 years, thus AE collection is up to three years starting from consent.
Description: Adverse events were not systematically collected for all subjects.
Arm/Group | Trental + Vitamin E
All-Cause Mortality (participants affected / at risk) | 15/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 4/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trental + Vitamin E (N=31)
Arrhythmia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Gait disturbance (General disorders) | 1 (1)
Generalized weakness (General disorders) | 1 (1)
Leg swelling (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Orthostatic dizziness (General disorders) | 1 (1)
Pain in shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Right leg weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Sleep disturbance (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT01508221/Prot_SAP_000.pdf